CLINICAL TRIAL: NCT02695095
Title: Comparison of the Risk of Acute Liver Injury Between Patients With Type 2 Diabetes Exposed to Dapafliglozin and Those Exposed to Other Antidiabetic Treatments
Brief Title: Acute Liver Injury in Patients on Dapagliflozin
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00005
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Acute Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To compare, by insulin use at the index date, the incidence of hospitalization for acute liver injury (ALI) among patients with type 2 diabetes mellitus who are new users of dapagliflozin with those who are new users of antidiabetic drugs (ADs) in classes other than sodium-glucose cotransporter 2 (SGLT2) inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylurea monotherapy.

DETAILED DESCRIPTION:
The overall goal of this research study is to estimate the risk of hospitalization for acute liver injury in patients who are prescribed dapagliflozin compared to patients prescribed other specific oral antidiabetic drugs. Dapagliflozin and other antidiabetic drugs are used to treat type 2 diabetes mellitus. Because of the mechanism of action for dapagliflozin and results from small safety monitoring studies, there is interest in further evaluating the safety of dapagliflozin in large populations.

The study will be implemented in three administrative health care data sources in two countries: in the United Kingdom, the Clinical Practice Research Datalink (CPRD); and in the United States, the Centers for Medicare and Medicaid Services (CMS) Medicare databases and the HealthCore Integrated Research Database (HIRDSM). Individuals in the databases will be included in the study if they meet the following age criteria; 18 years and older (CPRD and HIRD), or 65 years or older (Medicare); and if they did not have type 1 diabetes, are new users of one of the study drugs and meet the criteria of at least 180 days of electronic data before their first prescription of the study drug. The study period starts July 1, 2013 in CPRD, January 1, 2014 in PHARMO and January 9, 2014 in the United States data sources, and will end at the latest available data at each database at the time of analysis

ELIGIBILITY:
Inclusion Criteria:

1. receive newly prescribed dapagliflozin (with or without other ADs) or a newly prescribed AD (with or withoutother ADs) in a class other than SGLT2 inhibitors, insulin monotherapy, metformin monotherapy, or sulfonylureamonotherapy;
2. do not have evidence of type 1 diabetes;
3. are aged 18 years or older at the index date for CPRDpatients, 18-64 years for HIRDSM patients, or 65 years or older for Medicare patients; and
4. have been enrolled in the data source for at least 180 days before the first prescription or dispensing for dapagliflozin or comparator AD.

Exclusion Criteria:

* previous diagnosis of ALI; liver, biliary, or pancreatic disease; hepatobiliary or pancreatic neoplasm; or congestive heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are new users of dapagliflozin or the eligible comaprator drugs that meet the inclusion criteria and none of teh exclusion criteria.
  Comparator patients will be matched to the dapagliflozin patients by propensity score if access to all eligible comparator subjects is feasible.
Sampling Method: Non-Probability Sample
Enrollment: 424091 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
incidence of acute liver injury | Day after index day up to six years
  Patients will be followed from their index date (date of first study drug prescription or dispensing) until they experience one of the following: an event under study, end of time at risk for index medication, death, addition of a non-dapagliflozin (up to six years)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Johannes, Dr, Principal Investigator — RTI Health Solutions
Locations (3):
- United States (2):
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00005&attachmentIdentifier=b9cfda9c-42fa-4993-85f8-211004a2ec26&fileName=D1690R00005_CSR_Synopsis.pdf&versionIdentifier=